CLINICAL TRIAL: NCT03751475
Title: Optimized and Simplified Management of Acute Malnutrition in Children Aged 6 to 59 Months: a Community-based Clinical Randomized Controlled Trial in the Democratic Republic of Congo
Brief Title: Optimizing Acute Malnutrition Management in Children Aged 6 to 59 Months in Democratic Republic of Congo
Acronym: OptiMA-DRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for International Medical Action (Other)
Collaborators: Ministry of Public Health, Democratic Republic of the Congo (Other Government); The Innocent Foundation (Unknown); University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OptiMA-DRC
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Severe Acute Malnutrition; Moderate Acute Malnutrition; Child Malnutrition; Acute Malnutrition; Congo, The Democratic Republic of the; Africa; Randomized Clinical Trial
Keywords: Acute Malnutrition; Severe Acute Malnutrition; Moderate Acute Malnutrition; Child Malnutrition; Congo, The Democratic Republic of the; Randomized Clinical Trial; Africa
MeSH Terms: conditions — Severe Acute Malnutrition; Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: 2 parallel arms stratified on site and degree of acute malnutrition. 890 participants for the principal objective 480 participants with severe acute malnutrition for the secondary main objective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OptiMA (Experimental): The enrolled subjects will follow the nutritional Optima strategy.
  Interventions: Other: Nutritional Strategy - OptiMA
- Control (Active Comparator): The enrolled subjects will follow the standard nutritional protocol currently in use in the Democratic Republic of Congo
  Interventions: Other: Effective nutritional standard strategy

INTERVENTIONS:
Other: Nutritional Strategy - OptiMA — All children with a MUAC<125mm or oedema will be treated with the same RUTF, according to a new dosage table based on the evolution of MUAC and weight during recovery (RUTF dosage prescribed is gradually reduced as weight and MUAC increase).
  All children will be followed-up for 6 months following randomization. They will have weekly outpatient visit in the health facility until they meet discharge criteria, and then a bimonthly community-based follow-up in their villages (vital & anthropometric status and referral to the health facility for appropriate nutritional/medical care if indicated).
  Arms: OptiMA
Other: Effective nutritional standard strategy — Children presenting with MUAC<115 or WHZ<-3 or nutritional oedema, will be treated with RUTF, according to the usual dosage table based on weight at each visit.
  All children (whether eligible for RUTF or not) will be followed-up for 6 months following randomization. Children eligible for RUTF at randomization will have a weekly outpatient visit in the health facility until they meet discharge criteria, and then a bi-monthly community-based follow-up in their villages (vital & anthropometric status and referral to the health facility for appropriate nutritional/medical care if indicated). Children not eligible for RUTF at randomization will benefit from this same monthly community-based follow-up.
  Arms: Control

SUMMARY:
Acute malnutrition affects 51 million children under the age of 5 worldwide. Malnutrition contributes to nearly half of all child deaths each year, with the forms characterized by wasting or oedema (acute malnutrition) associated with the highest risk of death.

Although acute malnutrition is a continuum condition, it is arbitrarily divided into severe and moderate acute malnutrition (SAM, MAM) which are managed separately, with programs overseen by different UN agencies, and using different protocols and products. Such separation complicates delivery of care, contributes to high default and low coverage, and creates confusion among caregivers. Often treatment is only available for SAM children resulting in lives lost and costly hospitalisation that could be averted if nutritional support were available earlier in the wasting process. If we are to reduce the health and mortality burden from malnutrition, the effectiveness and cost-effectiveness of current protocols need dramatic improvements.

The dosage of Ready to Use Therapeutic Food (RUTF) for SAM (130-200 kcal/kg/d) has not changed since introduction of out-patient protocols in the mid-2000s. Children classified as SAM in these protocols are determined by three independent criteria: the presence of nutritional oedema or MUAC < 115 mm or weight-height Z score <-3. The RUTF dosage in these protocols is paradoxical in that the absolute amount of RUTF prescribed in the initial phases of treatment is often less than that given as the child nears recovery, because the number of packets in the weekly ration is determined by weight. However, rate of weight gain (g/kg/day) is highest in the first two weeks of treatment, and then plateaus - suggesting no benefit of increased RUTF amounts in the later phases of treatment. Progressive reduction seems to be a more rational use of RUTF.

The Optimizing treatment for acute MAlnutrition (OptiMA) strategy consists in simplifying management of acute malnutrition through the use of a single anthropometric admission criterion (mid upper arm circumference [MUAC] < 125 mm or nutritional oedema) - one that best captures children's anthropometry related mortality risk- and by optimizing the use of RUTF by adapting doses to the nutritional recovery of the child. RUTF doses begin at 170 kcal/kg/d for the most severely wasted (MUAC < 115 mm or oedema) and reduce to 75 kcal/kg/d as oedema resolves and MUAC increases > 120 mm.

The investigators hypothesize that this strategy could double the number of children in care compared to current SAM programs without substantially increasing the amount of RUTF or staffing required while maintaining a recovery rate in line with current programs. OptiMA may also improve coverage and reduce the need for hospitalization through early identification of malnourished children.

The investigators propose to conduct a community-based non-inferiority clinical trial with individual randomization comparing the OptiMA strategy to the Democratic Republic of Congo standard nutritional protocol for SAM. Study children will be randomly assigned to the intervention arm or control arm - with children at MUAC < 125 mm or oedema eligible for RUTF in the intervention arm and those meeting current WHO SAM definition eligible in the control group. All participants will be followed for 9 months post-randomization to assess non-inferiority as defined by a composite of three endpoints : alive, acceptable nutritional status (MUAC ≥ 125 mm and WHZ >-3, no oedema) and no relapse to acute malnutrition for those who were treated with RUTF. The main secondary outcome will assess the non-inferiority of OptiMA RUTF dosing (170 kcal/kg/d) in children meeting current WHO SAM criteria compared to children with the same criteria in the control arm who will receive 130-200 kcal/kg/d.

DETAILED DESCRIPTION:
The OptiMA strategy proposes a new malnutrition management approach, grounded in 3 main principles.

Firstly, the diagnosis of acute malnutrition is refined to target those at highest mortality risk within the CMAM definition of acute malnutrition (WHZ < -2 or MUAC < 125 mm or oedema), by targeting treatment to children with a MUAC < 125 mm or oedema. The simplicity of MUAC measure allows families to screen children and check for oedema at home and identify malnourished children at an earlier stage. The diagnosis is quickly confirmed by clinicians at the health center. MUAC progression is also used to monitor recovery and determine discharge thus eliminating the discrepancies that occur when both MUAC and WHZ are used to diagnose acute malnutrition.

Secondly, RUTF dosage is rationalized, and calibrated to the child's degree of wasting. The WHZ tables and dosing tables are replaced by a single table that determines the child's RUTF ration based on MUAC category and weight. Larger rations, on a per kilo basis, are given to the most severely malnourished and the ration is reduced as the child progresses to recovery.

Thirdly, supply chain is simplified to a single RUTF and data management from 2 programs are merged into one. This streamlined programme should result in better coverage, a high proportion of children detected before MUAC<115 mm, lower RUTF consumption per child and fewer acute malnutrition related hospitalisations.

ELIGIBILITY:
Inclusion Criteria:

* Be between 6 and 59 months old;
* Meet one of the acute malnutrition criteria defined as follows: PB < 125mm or ratio Weight/Size (Z-score) <-3 (WHO standard) or Oedema of grade +, ++;
* Be resident in the health area where the active screening session takes place;
* Have the free, informed and signed consent of the child's mother or guardian.

Exclusion Criteria:

* Children with medical complication or negative appetite test or oedema (grade +++)
* Children allergic to milk or peanuts;
* Children suffering from a known chronic pathology such as sickle cell anemia, trisomy 21, congenital heart disease, or neurological condition;
* Children currently in a malnutrition programme.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 896 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Success rate in each arm | 6 months after randomization
  Success is defined by a composite indicator evaluated 6 months post-randomization:
  * child alive and not acutely malnourished, per the same definition at inclusion : absence of oedema and MUAC ≥125mm and WHZ ≥-3 and
  * for the duration of the 6-month observation period following randomization, the child does not develop another episode of acute malnutrition applying the same definition at study inclusion.

SECONDARY OUTCOMES:
Recovery rate in participants with severe acute malnutrition (WHO definition) | After RUTF treatment, through the 6 month study completion
  The recovery rate is defined by a MUAC≥125 (OptiMA arm) and a MUAC≥125 or a WHZ>-1.5 (Standard Protocol arm) during two consecutive visits, absence of oedema, minimum treatment period of 4 weeks and good clinical condition

OTHER OUTCOMES:
Consumption of RUTF | At the visit of recovery status occuring through the 6 month study completion
  Comparaison of the median/mean of the total number of RUTF sachet administred between both arms in recovered SAM
Total weight gain and daily weight gain | At the visit of recovery status occuring through the 6 month study completion
  Comparaison of the median/mean of the total weight gain in grams and the daily weight gain in g/kg/d between both arms in recovered SAM children
Total MUAC gain and daily MUAC gain | At the visit of recovery status occuring through the 6 month study completion
  Comparaison of the median/mean of the total MUAC gain in mm and of the MUAC gain in mm/day in recovered SAM children between both arms
Total length of RUTF treatment | At the visit of recovery status occuring through the 6 month study completion
  Comparaison of the median/mean of the total number of days with RUTF treatment in recovered SAM children between both arms.
Absence of recovery | After 12 and after 16 weeks of nutritional follow-up
  Comparaison of the proportion of absence of recovery in SAM children at inclusion between both arms
Mortality | Through the 6 month study completion
  Comparaison of the death proportion in children with AM at inclusion and in children with SAM at inclusion between both arms in each population
Hospitalisation | Through the 6 month study completion
  Comparaison of the proportion of hospitalisation in children with AM at inclusion and in children with SAM at inclusion between both arms in each population
Relapse to a new episode of AM and to a new episode of SAM | During a 3 months period following the recovered episode of AM or of SAM at inclusion
  Comparaison of the proportion of children who relapse to a new episode of AM and to a new episode of SAM in SAM children at inclusion and in children with AM at inclusion between both arms in each population

CONTACTS AND LOCATIONS:
Overall Officials: SHEPHERD SUSAN, MD, Principal Investigator — Alliance for International Medical Action; BECQUET RENAUD, MPH, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Health Zone, Kamuesha, Kasai Province, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
The research findings will be disseminated in peer-reviewed journals, meetings and international conferences.
  Individual participant data will be accessible through controlled access repositories, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: SAP : before end of the study on ClinicalTrials.gov Individual participant data : Beginning 6 months and ending 36 months following article publication. After 36 months the data will be available in our University's data warehouse and in co-investigators (Programme National Nutrition of DRC) data warehouse.
Access Criteria: Study Protocol and ICF(both in french) can be shared on request Individual participant data : researchers who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee

REFERENCES:
- [Background] Cazes C, Phelan K, Hubert V, Alitanou R, Boubacar H, Izie Bozama L, Tshibangu Sakubu G, Beuscart A, Yao C, Gabillard D, Kinda M, Augier A, Anglaret X, Shepherd S, Becquet R. Simplifying and optimising management of acute malnutrition in children aged 6 to 59 months: study protocol for a community-based individually randomised controlled trial in Kasai, Democratic Republic of Congo. BMJ Open. 2020 Dec 2;10(12):e041213. doi: 10.1136/bmjopen-2020-041213. PMID 33268424
- [Result] Cazes C, Phelan K, Hubert V, Boubacar H, Bozama LI, Sakubu GT, Tshiala BK, Tusuku T, Alitanou R, Kouame A, Yao C, Gabillard D, Kinda M, Daures M, Augier A, Anglaret X, Shepherd S, Becquet R. Simplifying and optimising the management of uncomplicated acute malnutrition in children aged 6-59 months in the Democratic Republic of the Congo (OptiMA-DRC): a non-inferiority, randomised controlled trial. Lancet Glob Health. 2022 Apr;10(4):e510-e520. doi: 10.1016/S2214-109X(22)00041-9. PMID 35303461
- [Result] Cazes C, Phelan K, Hubert V, Boubacar H, Bozama LI, Sakubu GT, Senge BB, Baya N, Alitanou R, Kouame A, Yao C, Gabillard D, Daures M, Augier A, Anglaret X, Kinda M, Shepherd S, Becquet R. Optimising the dosage of ready-to-use therapeutic food in children with uncomplicated severe acute malnutrition in the Democratic Republic of the Congo: a non-inferiority, randomised controlled trial. EClinicalMedicine. 2023 Feb 28;58:101878. doi: 10.1016/j.eclinm.2023.101878. eCollection 2023 Apr. PMID 36915287
- [Derived] Hubert V, Phelan K, Bozama LI, Boubacar H, Sakubu GT, Tshiala B, Savy M, Becquet R, Cazes C. Food insecurity, feeding practices and associated factors of acute malnutrition among children under 5 years of age in a post-conflict context in the Kasai region, Democratic Republic of Congo: a community-based case-control study. BMC Nutr. 2025 May 30;11(1):106. doi: 10.1186/s40795-025-01096-0. PMID 40448235